CLINICAL TRIAL: NCT02762591
Title: Expanded Access Program of Pimavanserin in Patients With Parkinson's Disease Psychosis
Brief Title: Expanded Access of Pimavanserin for Patients With PD Psychosis
Status: Approved for marketing | Type: Expanded Access
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ACP-103-036
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Parkinson's Disease Psychosis
MeSH Terms: interventions — pimavanserin

INTERVENTIONS:
Drug: Pimavanserin tartrate — Pimavanserin tartrate 40 mg, tablet, taken as two 20 mg tablets, once daily by mouth

SUMMARY:
The purpose of this program is to provide patients with PDP access to pimavanserin until the product receives marketing approval from the FDA and is commercially available.

ELIGIBILITY:
Inclusion Criteria:

1. Patient meets one of the following criteria:

   1. Patient has participated in a previous study of pimavanserin for Parkinson's disease psychosis (PDP)
   2. New ("De novo") patients
2. A clinical diagnosis of Parkinson's disease with a minimum duration of 1 year
3. Female patients must be of non-childbearing potential
4. Psychotic symptoms must have developed after Parkinson's disease diagnosis was established
5. Patient that has received stereotaxic surgery for subthalamic nucleus deep brain stimulation must be at least 6 months post-surgery and the stimulator settings must have been stable for at least 1 month prior to Study Day 1 (Baseline) and must remain stable during the trial
6. The patient or Legally Authorized Representative (LAR) is willing and able to provide consent
7. The patient or LAR is willing and able to adequately communicate in English.

Exclusion Criteria:

1. Patient has a history of significant psychotic disorders prior to or concomitantly with the diagnosis of Parkinson's disease including, but not limited to, schizophrenia or bipolar disorder
2. Patient has had dementia prior to or concurrently with their diagnosis of Parkinson's disease that may be inconsistent with a Parkinson's diagnosis
3. Patient has current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, renal, hematologic, or other medical disorder, including cancer or malignancies, which would affect the patient's ability to participate in the program
4. Patient has had a myocardial infarction in last six months
5. Patient has any surgery planned during the screening, treatment, or follow-up periods

Patients will be evaluated at screening to ensure that all criteria for study participation are met. These evaluations will include specific measures of psychosis severity, delirium, dementia, cardiovascular condition, and pregnancy status. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult